CLINICAL TRIAL: NCT02879734
Title: Comparison Between Performing Prophylactic Omentopexy and Lack of Omentopexy During Laparoscopic Insertion of Peritoneal Dialysis Catheters in Terms of Complications and Catheter Function
Brief Title: Prophylactic Omentopexy During Laparoscopic Insertion of Peritoneal Dialysis Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IR.TUMS.VCR.REC.1395.247
Record Dates: First submitted 2016-08-04; First posted 2016-08-26 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2016-08

CONDITIONS: Mechanical Complication of Peritoneal Dialysis Catheter
Keywords: peritoneal dialysis; laparoscopy; omentum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without Omentopexy (No Intervention): Patients that did not undergo prophylactic omentopexy during laparoscopic insertion of peritoneal dialysis catheter
- With Omentopexy (Experimental): Patients that underwent prophylactic omentopexy during laparoscopic insertion of peritoneal dialysis catheter. Intervention = Prophylactic laparoscopic omentopexy
  Interventions: Other: Prophylactic laparoscopic omentopexy

INTERVENTIONS:
Other: Prophylactic laparoscopic omentopexy — Fixation of omentum with sutures to anterior abdominal wall during laparoscopic surgery
  Arms: With Omentopexy

SUMMARY:
The purpose of this study is to compare function of the peritoneal dialysis catheter in two groups of patients with and without prophylactic omentopexy that was performed during laparoscopic insertion of peritoneal catheters.

DETAILED DESCRIPTION:
Peritoneal dialysis is a know and accepted treatment in patients with end stage renal diseases. The is a safe, easy and cheap treatment modality in these patients. After introduction and development of laparoscopic procedures for insertion of peritoneal dialysis catheters, some prophylactic surgical techniques have been proposed as measures to reduce catheter malfunction. Omentopexy is among these techniques. The purpose of this study is to compare function of the peritoneal dialysis catheter (including inflow and outflow failure) in two groups of patients with and without prophylactic omentopexy that was performed during laparoscopic insertion of peritoneal catheters.

ELIGIBILITY:
Inclusion Criteria:

• End-stage renal failure in need of prolonged dialysis referred for insertion of peritoneal dialysis catheter

Exclusion Criteria:

* Contraindications to laparoscopic surgery
* Coagulative disorder
* Death of participant due to other reasons before usage of peritoneal catheter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Ability of the peritoneal catheter to pass the dialysis fluid | One months
  Inflow and outflow passage of the peritoneal dialysis fluid from the catheter based on questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Reza Keramati, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Mohammad Reza Keramati, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No